CLINICAL TRIAL: NCT07365111
Title: Insights Into the Characteristics, Prescription and Delivery of Continuous Renal Replacement Therapy to Critical Ill Patients - The iCRRT Data Registry
Brief Title: Insights Into the Continuous Renal Replacement Therapy to Critical Ill Patients
Acronym: iCRRT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Zagreb (Other)
Responsible Party: Principal Investigator, Oleksa Rewa, Associate Professor, Director of Research & Innovation, University of Alberta
Other Study IDs: Pro00160785
Record Dates: First submitted 2025-12-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Continuous Renal Replacement Therapy (CRRT); Acute Kidney Injury; Renal Dialysis; Critical Illness
Keywords: Continue Renal Replacement Therapy; Dialysis; Acute Kidney Injury; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Any patients admitted to the ICU and required CRRT
  Interventions: Device: continuous renal replacement therapy

INTERVENTIONS:
Device: continuous renal replacement therapy — We will include any critically ill patient admitted to an intensive care unit requiring dialysis
  Other Names: CRRT

SUMMARY:
This is a multinational, prospective, observational study designed to characterize patient demographics, prescription parameters, and process measures of continuous renal replacement therapy (CRRT) in intensive care units (ICUs) worldwide. The study aims to examine similarities and differences in CRRT practices and outcomes among critically ill adult patients across a global network of medical centers.

The goal is to develop a large, comprehensive repository of data on CRRT practices and outcomes. This repository will enable characterization of variation in standard CRRT practices across medical centers. Natural variability in practice patterns-both between and within centers-will provide an opportunity to compare outcomes associated with different approaches and to generate high-quality preliminary data to inform future interventional trials.

Primary Objective

- To describe global patient characteristics, CRRT modalities, and clinical outcomes among patients receiving CRRT.

Secondary Objectives

* To compare clinical outcomes across geographic regions and CRRT modalities.
* To identify patient-level and practice-level predictors of outcomes.
* To assess the impact of comorbid conditions (e.g., diabetes mellitus) on CRRT outcomes.

Exploratory Objectives

* To evaluate long-term renal outcomes and patient-reported quality of life.
* To explore health economics and resource utilization related to CRRT.

Study Population All patients receiving CRRT as part of routine clinical care in the ICU at participating centers will be eligible for inclusion.

Data Collection The study will support an epidemiological assessment of patients undergoing CRRT, including, but not limited to, demographics, underlying disease states, severity of illness, physiological support, indications for CRRT, and clinical outcomes. Outcomes of interest include ICU and hospital mortality, ICU and hospital length of stay, and renal recovery.

DETAILED DESCRIPTION:
1.0 Rationale The goal of this study is to develop a large repository of data on CRRT practices and outcomes, enabling characterization of similarities and differences in standard CRRT practices across medical centers. Natural variability in practices will provide an opportunity to compare outcomes associated with different practice patterns and generate important preliminary data to inform future interventional trials.

2.0 Background Despite the accumulation of high-quality evidence, the prescription, delivery, and maintenance of continuous renal replacement therapy (CRRT) remain highly variable across clinical settings. This persistent heterogeneity reflects uncertainty in key aspects of CRRT practice and underscores the need for a comprehensive, international evaluation. The international CRRT (iCRRT) initiative was established to systematically characterize global CRRT practices, identify regional variation, and inform strategies to optimize the delivery of this life-sustaining therapy for critically ill patients.

Acute kidney injury (AKI) is among the most common and severe complications encountered in critical illness, affecting more than half of patients admitted to intensive care units (ICUs). Approximately 6% of ICU patients require renal replacement therapy (RRT), a subgroup in whom hospital mortality remains exceedingly high, frequently approaching or exceeding 50%. Although AKI is associated with substantial morbidity, mortality, and healthcare utilization, no interventions have been shown to consistently reverse established kidney injury. Management, therefore, remains largely supportive, with RRT reserved for patients with advanced or refractory disease.

For critically ill patients, particularly those with hemodynamic instability, CRRT has become the predominant RRT modality in many high-income countries. Since the original description of continuous arteriovenous hemofiltration more than three decades ago, technological and procedural advances have transformed CRRT into a widely adopted and routinely applied therapy. Compared with intermittent hemodialysis (IHD), CRRT offers superior hemodynamic tolerance, continuous solute control, and more precise fluid management. These perceived advantages form the basis of the 2012 Kidney Disease Improving Global Outcomes (KDIGO) guidelines, which recommend CRRT over intermittent modalities in hemodynamically unstable patients . Nevertheless, despite its central role in contemporary critical care, substantial variation in CRRT practice persists across institutions and individual providers.

At the same time, there is increasing recognition that traditional clinical outcomes alone may incompletely capture the impact of critical illness and its treatments. Evidence increasingly supports the routine use of patient-reported outcome measures (PROMs) to improve patient-clinician communication, enhance patient satisfaction, and positively influence health-related quality of life (HRQL). In this context, the Alberta-based EMPATHY study is evaluating the effectiveness and cost-effectiveness of systematic PROMs collection in chronic RRT programs, examining associations with patient experience, clinical outcomes, HRQL, and healthcare utilization.

Despite existing guideline recommendations-most notably regarding target effluent dose and the preferential use of regional citrate anticoagulation - guidance remains limited for many fundamental components of CRRT delivery, including modality selection, anticoagulation protocols, electrolyte supplementation, and fluid balance strategies. This lack of consensus reflects the limited strength of the current evidence base, which is largely derived from small, single-center studies. Moreover, despite the high-risk nature of patients receiving CRRT, quality indicators and patient safety outcomes related to CRRT delivery have been insufficiently studied.

In this context, the investigators describe the protocol for a prospective observational study designed to evaluate CRRT practices among critically ill adult patients across an international consortium of medical centers. The primary objective is to establish a large, multicenter repository capturing patient characteristics, CRRT prescription and delivery patterns, and associated clinical outcomes. By leveraging natural variation in practice across healthcare systems, this study aims to generate robust comparative data and provide a foundation for the design of future interventional trials aimed at improving CRRT care and outcomes worldwide.

3.0 Research Question What are the similarities and differences in CRRT practices and outcomes among critically ill adult patients across a network of global medical centres?

4.0 Objectives Primary Objective

-To describe global patient characteristics, CRRT modalities, and clinical outcomes among patients receiving CRRT.

Secondary Objectives

* To compare outcomes across geographic regions and CRRT modalities.
* To identify patient-level and practice-level predictors of outcomes.
* To assess the impact of comorbidities (e.g., diabetes mellitus, chronic obstructive pulmonary disease, cerebrovascular accidents and hypertension) on CRRT outcomes.

Exploratory Objectives

* To evaluate long-term renal outcomes and quality of life.
* To explore health economics and resource utilization related to CRRT.

5.0 Methods Design and Setting This is a multinational, prospective, observational study designed to characterize patient demographics, prescription parameters, and process measures of continuous renal replacement therapy (CRRT) in intensive care units (ICUs) worldwide.

Study Population The study will be conducted in ICUs at participating centers globally. All critically ill patients receiving CRRT as part of routine ICU care will be eligible for inclusion. Inclusion criteria are intentionally broad to capture a systems-level population suitable for evaluating practice patterns and outcomes.

Inclusion Criteria

* Admission to the ICU
* Receipt of CRRT therapy Exclusion Criteria
* End-stage kindey disease
* CRRT < 24 hours

Sample Size No formal sample size calculation will be performed. All eligible patients will be included.

Interventions CRRT administered as part of routine ICU care. This is an observational study; no study-related clinical interventions will be performed, and no biospecimens will be collected.

Data Collection A comprehensive range of data will be collected, including patient characteristics at enrolment, CRRT modalities and treatment courses, fluid balance, medications, and clinical outcomes. Electronic medical records will serve as the primary data source.

Each site will assign a de-identified patient identification number through the registry database; no direct patient identifiers will be uploaded. Sites without electronic medical records may manually enter de-identified data into a secure, password-protected, web-based interface. All electronic data transmission will use encryption technology to ensure data privacy and security.

The registry will comply with applicable privacy regulations, including the Health Insurance Portability and Accountability Act (HIPAA; 45 CFR Parts 160 and 164), including provisions related to de-identified data and limited data sets.

All sites will use standardized electronic case report forms. Measurement units will be customized to reflect local laboratory reporting practices, with automatic conversion and storage of values in standardized units for centralized analysis.

Statistical Analysis Data will be summarized using standard descriptive statistical methods. Associations between patient characteristics, CRRT initiation and prescription parameters, and clinical outcomes (including mortality, length of stay, and duration of AKI) will be evaluated using analysis of variance (ANOVA) for normally distributed variables or the Kruskal-Wallis test for non-normally distributed variables. Multivariable models will be developed, including variables with a univariate significance level of p < 0.20 and/or based on clinical relevance as determined by investigators judgment. Additional analyses will be conducted to address specific research questions as they arise.

Primary Outcomes An epidemiological assessment of patients undergoing CRRT, including, but not limited to, demographics, disease states, severity of illness, physiological support, indications for CRRT, and clinical outcomes. Outcomes include ICU and hospital mortality, ICU and hospital length of stay, and renal recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to an intensive care unit
2. CRRT therapy

Exclusion Criteria:

1. End-stage kidney disease
2. CRRT <24 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with new acute kidney injury and initiation of continuous renal replacement therapy who are admitted to an intensive care unit and who have received continuous renal replacement therapy for at least 24 hours will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2036-03-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 28 days
  Patient survival at the time of ICU discharge

SECONDARY OUTCOMES:
Hospital mortality | Up to 90 days
  Patient survival status during their hospitalization
ICU length of stay | Up to 90 days
  Duration of ICU stay
Hospital length of Stay | Up to 90 days
  Duration of hospital stay
Renal recovery | Up to 90 days
  1) Return of serum creatinine (SCr) to within 50% of baseline; 2) no longer receiving dialysis
Adverse events | Up to 90 days
  Any adverse events adjudicated to CRRT-related events

OTHER OUTCOMES:
Health Related Quality of Life | 90 and 365 days
  Health Related Quality of Life (EQ-5D-5L) "EuroQol 5-Dimension 5-Level" questionnaire.
Health Economic Analysis | Up to 90 days
  ICU and Hospital Costs

CONTACTS AND LOCATIONS:
Overall Officials: Oleksa Rewa, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided